CLINICAL TRIAL: NCT01863446
Title: Effects of Light on Melatonin and Contractions in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Harvard University (Other); National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Elizabeth Klerman MD PhD, Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2012P002568; 1R21HD086392-01 (NIH)
Record Dates: First submitted 2013-05-23; First posted 2013-05-29 (Estimated); Results first posted 2023-11-13 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Pregnancy
Keywords: Pregnancy; Melatonin; Contractions; Light

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Lighting1 (Experimental): Ocular light exposure of a red wavelength light for one night
  Interventions: Device: Lighting1
- Lighting2 (Experimental): Ocular light exposure of a blue-green wavelength light for one night
  Interventions: Device: Lighting2
- Lighting3 (Experimental): Ocular light exposure to a red wavelength light on night 1 and to a red wavelength light on night 2
  Interventions: Device: Lighting1
- Lighting4 (Experimental): Ocular light exposure to a red wavelength light on night 1 and to a blue-green wavelength light on night 2
  Interventions: Device: Lighting1; Device: Lighting2

INTERVENTIONS:
Device: Lighting1 — Ocular light exposure to a red wavelength light
  Arms: Lighting1; Lighting3; Lighting4
Device: Lighting2 — Ocular light exposure to a blue/green wavelength light
  Arms: Lighting2; Lighting4

SUMMARY:
Specific Aim: Test the hypothesis that ocular light exposure will suppress melatonin secretion and reduce uterine contractions in women at late term pregnancies.

Secondary aim. Test the hypothesis that ocular light exposure will reduce self-reported uterine contractions in women at late term pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* pregnant at 35-40 weeks
* first pregnancy

Exclusion Criteria:

* pregnancy-related complications
* twin or higher pregnancy
* using medication that affects the sympathetic nervous system

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2013-05; Primary Completion 2021-06 (Actual); Study Completion 2023-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth B Klerman, MD PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 51 people total enrolled 33 started study; 18 were not studied. 18 people who signed informed consent were not studied: 3 had a new medical reason for ineligibility 5 delivered the baby before their scheduled study date 8 signed consent forms but were not studied because study enrollment was complete before their scheduled study data 2 were lost to follow-up
Groups:
- Lighting4: Ocular light exposure to a red wavelength light on night 1 and to a blue-green wavelength light on night 2
  Lighting1: Ocular light exposure to a red wavelength light Lighting 2: Ocular light exposure to a blue/green wavelength light
Period: Overall Study
Arm/Group | Lighting1 | Lighting2 | Lighting3 | Lighting4
Started | 5 | 4 | 12 | 12
Completed | 4 | 4 | 10 | 10
Not Completed | 1 | 0 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 2
Not completed — Physician Decision | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Incomplete data (problem with data collection) in 2 participants in Lighting 3 and 1participant in Lighting4
Groups:
- Total: Total of all reporting groups
Arm/Group | Lighting1 | Lighting2 | Lighting3 | Lighting4 | Total
Number analyzed (Participants) | 4 | 4 | 8 | 9 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] — Age, Continuous in years
  years | 24.8 (5.4) | 23.0 (4.7) | 27.5 (4.9) | 30.4 (3.2) | 27.4 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8 | 9 | 25
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 2 | 6
  Not Hispanic or Latino | 3 | 3 | 6 | 7 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 1 | 3 | 2 | 1 | 7
  White | 2 | 1 | 5 | 7 | 15
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Gestational age [Mean (Standard Deviation); unit: weeks] — Population: data are missing about gestational age for three participants
  weeks
    number analyzed (Participants) | 4 | 4 | 6 | 8 | 22
    (all) | 37.9 (1.2) | 37.6 (1.2) | 38.3 (0.4) | 37.7 (1.1) | 37.9 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Melatonin Area Under the Curve (AUC)
Description: Melatonin will be assessed using concentrations in saliva or blood. AUC will be calculated using melatonin concentrations during the Outcome Measure Time Frame.
  (1) for Lighting1 and Lighting2, the AUC for night 1; (2) for Lighting3 and Lighting4, the AUC for Night 2
Time Frame: 4 hours of light exposure.
Population: Healthy pregnant women. In Lighting3, there were missing data from 2 participants; in Lighting4, there were missing data from 1 participant
Measure: Mean (Standard Deviation); unit: area under curve (h*pg/mL)
Arm/Group | Lighting1 | Lighting2 | Lighting3 | Lighting4
Number analyzed (Participants) | 4 | 4 | 8 | 9
area under curve (h*pg/mL) | 42.1 (23.0) | 24.3 (24.8) | 38.5 (14.6) | 26.3 (39.8)
Statistical Analysis 1: Comparison: Lighting1 vs Lighting2; Test type: Superiority — Unpaired t-test comparing Lighting 1 and Lighting2; p = 0.334, t-test, 2 sided
Statistical Analysis 2: Comparison: Lighting3 vs Lighting4; Test type: Superiority — Unpaired t-test comparing Lighting3 vs Lighting 4; p = 0.423, t-test, 2 sided

2. Secondary Outcome: Uterine Contractions
Description: Uterine contractions will be measured using a uterine tocometer device
  (1) for Lighting1 and Lighting2, the sum for night 1; (2) for Lighting3 and Lighting4, the sum for Night 2
Time Frame: 4 hours of light exposure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of uterine contractions
Arm/Group | Lighting1 | Lighting2 | Lighting3 | Lighting4
Number analyzed (Participants) | 4 | 4 | 8 | 9
number of uterine contractions | 16.8 (10.9) | 13.8 (17.3) | 14.5 (9.1) | 13.0 (12.8)
Statistical Analysis 1: Comparison: Lighting1 vs Lighting2; Test type: Superiority — Unpaired t-test of Lighting1 vs Lighting2; p = 0.780, t-test, 2 sided
Statistical Analysis 2: Comparison: Lighting3 vs Lighting4; Test type: Superiority — Unpaired t-test of Lighting3 vs Lighting4; p = 0.791, t-test, 2 sided

3. Other Pre Specified Outcome: Subjective Assessment of Uterine Contractions
Description: Self-reported uterine contractions will be assessed by asking the women how many contractions they felt.
  (1) for Lighting1 and Lighting2, the sum for night 1; (2) for Lighting3 and Lighting4, the sum for Night 2
Time Frame: 4 hours of light exposure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of uterine contractions
Arm/Group | Lighting1 | Lighting2 | Lighting3 | Lighting4
Number analyzed (Participants) | 4 | 4 | 8 | 9
number of uterine contractions | 4.0 (6.1) | 3.5 (2.4) | 5.5 (4.9) | 2.9 (4.5)
Statistical Analysis 1: Comparison: Lighting1 vs Lighting2; Test type: Superiority — Unpaired t-test; p = 0.883, t-test, 2 sided
Statistical Analysis 2: Comparison: Lighting3 vs Lighting4; Test type: Superiority — Unpaired t-test; p = 0.271, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Inpatient 1 or 2 days
Arm/Group | Lighting1 | Lighting2 | Lighting3 | Lighting4
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-10-18): https://cdn.clinicaltrials.gov/large-docs/46/NCT01863446/Prot_SAP_ICF_000.pdf